CLINICAL TRIAL: NCT02962817
Title: The Influence of an Educational Internet-based Intervention in the Beliefs and Attitudes of Primary Care Professionals on Non-specific Chronic Low Back Pain: Study Protocol of a Mixed Methods Approach
Brief Title: The Influence of an Educational Intervention in the Beliefs and Attitudes of Primary Care Professionals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Ester García Martínez, Ester García Martínez, Faculty of Nursing and Physiotherapy, Universitat de Lleida, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ULleida P16/124
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Chronic Nonspecific Low Back Pain
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational intervention through a web platform (Experimental): This group will have access to our web platform where they will find information related to nonspecific chronic low back pain. This information will be presented through dynamic explanatory 3D videos made by the author.
  The aim of this intervention is to change and modify wrong beliefs and attitudes about chronic low back pain of physicians and nurses working in primary care settings, using a web-based educational tool with the additional result of increasing knowledge on pain neurophysiology and reducing fear-avoidance beliefs.
  Interventions: Other: Educational intervention
- Clinical practice guidelines on low back pain (Active Comparator): Control group: They will have access to a video where medical staff and primary care nurses explain the content of the clinical practice guideline for addressing back pain.
  Interventions: Other: Video explaining the clinical practice guidelines on low back pain

INTERVENTIONS:
Other: Educational intervention
  Arms: Educational intervention through a web platform
Other: Video explaining the clinical practice guidelines on low back pain
  Arms: Clinical practice guidelines on low back pain

SUMMARY:
Aim: The primary aim of this project is to identify the fear-avoidance beliefs and attitudes of primary care physicians and nurses towards the treatment of chronic nonspecific low back pain to subsequently develop a biopsychosocial educational tool using a web platform. The secondary aim of this project is to evaluate the effectiveness of this educational intervention about pain neurophysiology and fear-avoidance beliefs, using a web platform for primary care physicians and nurses.

Methods: Exploratory sequential mixed method design. For the qualitative phase of this study, researchers will use personal semistructured interviews. For the quantitative phase the authors will use an experimental study design.

Subjects: medical and nursing staff working in primary care centers in the city of Lleida, Spain.

Expected outcomes: the authors expect to change and modify wrong beliefs and attitudes about chronic low back pain of physicians and nurses working in primary care settings, using a web-based educational tool with the additional result of increasing knowledge on pain neurophysiology and reducing fear-avoidance beliefs.

DETAILED DESCRIPTION:
HYPOTHESIS AND OUTCOMES

Hypothesis:

1. The beliefs and attitudes of fear-avoidance of primary care professionals are held by lack of knowledge about the origin and meaning of pain.
2. The neurophysiology of pain as a biopsychosocial educational intervention using a web platform for primary care professionals will change their knowledge about the origin and meaning of pain, with the result of reducing the beliefs and attitudes of fear avoidance.

Outcomes:

* Qualitative:

  1. To identify the fear-avoidance beliefs and attitudes of primary care professionals towards the treatment of chronic nonspecific low back pain in relation to the origin and meaning of pain.
  2. To build and develop using a web platform a biopsychosocial educational intervention based on the results obtained in the qualitative phase.
* Quantitative:

  1. To evaluate the effectiveness of a biopsychosocial educational intervention about pain neurophysiology and fear-avoidance beliefs related to non-specific chronic low back pain, using a web platform for primary care professionals.

METHODOLOGY DESING To answer the research question a mixted-method sequential exploratory design will be used. This mixed-method design consists of two stages, where the results of the methodology used in the first phase of the study, in this case qualitative, contribute to the development of the second quantitative phase. In this project, both phases should have the same relevance for the development of an educational tool for primary care professionals. Using a mixed design methodology is justified in this protocol because the integration of both (qualitative and quantitative) methodologies occurs when data from the qualitative phase contributes to the construction of an educational tool.

The process to be followed is:

* Qualitative: Semistructured personal interviews.
* Quantitative: An experimental study design in which a sample of specialized physicians in family and community care and nurses working in primary care health centers will be randomly assigned to the experimental group and the control group.

SUBJECTS:

- Qualitative and quantitative: To start the recruitment process, the principal investigator will do a presentation of the project in each of the primary care centers in the city of Lleida addressed to the medical and nursing staff. Professionals will be invited to participate in the study, either in the qualitative or quantitative phase, and will be provided a phone number and an email address through which they can contact the researcher and agree on the interview date. In the quantitative phase, health professionals who meet the inclusion criteria will be informed about the intervention and the author will answer any questions or concerns that may arise. At the end of this first contact the professionals will be asked to read and sign the informed consent.

* Qualitative: Subjects who agree to be part of the qualitative study will be contacted by the author and invited to participate in a deep semistructured interview. Individual interviews will be conducted in Spanish or Catalan and will be audio recorded with the consent of interviewed professionals. To increase participation, interviews will be conducted in designated areas in the primary health centers, during working hours. The duration of the interview will be approximately 1 hour.
* Quantitative: Subjects will be randomly allocated to either intervention or control group using a simple randomization method.

Intervention group: This group will have access to the web platform where they will find information related to nonspecific chronic low back pain. This information will be presented using dynamic explanatory videos made by the author.

Control group: They will have access to a video where medical staff and primary care nurses explain the content of the clinical practice guidelines for addressing back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Graduated in medicine and specialized in family and community medicine.
2. Graduates in nursing.
3. Registered health professionals.
4. Professionals working in any of the primary care centers.
5. Accept and sign the informed consent form.

Exclusion Criteria: nothing

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-02 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Knowledge about the pain neurophysiology | 2 weeks
  Using the pain neurophysiology questionnaire. This self-administered questionnaire was developed by Lorimer Moseley in 2003 to assess how an individual conceptualizes pain. An acceptable internal consistency and good test-retest reliability was demonstrated. The original English version was translated into Spanish by the Language Service of the Rovira and Virgili University. The questionnaire consists of 19 statements that refer to the origin and meaning of pain with three possible answers: true, false or doubtful. Each correct answer is scored with 1 point, while incorrect, doubtful or unanswered responses are scored with 0 points.

SECONDARY OUTCOMES:
Fear-avoidance beliefs | 2 weeks
  Using the Health Care Providers Pain and Impairment Relationship Scale. This self-administered questionnaire was designed to assess attitudes and beliefs of primary care physicians on chronic nonspecific low back pain. Domenech et al. translated into Spanish the original English version in 2013. After the cross-cultural adaptation, the Spanish version of HC-PAIRS proved to be a reliable, valid and sensitive instrument. The questionnaire consists of 15 statements that suggest a direct link between pain and functional limitation and disability. Each statement is followed by a 7 point Likert scale (1 = strongly disagree, 4 = neither agree nor disagree and 7 = strongly agree). The total score ranges from 1 to 105. Higher scores indicate strong beliefs.
Fear-avoidance beliefs and attitudes | 2 weeks
  Using the Fear Avoidance Beliefs Questionnaire. This self-administered questionnaire was developed to measure the beliefs and attitudes of fear-avoidance in patients with low back pain towards physical and / or occupational activities. The questionnaire is divided into two subscales: FABQ-physical activity and FABQ-work. It consists of a total of 16 statements about the beliefs of patients with low back pain about the relationship between pain and physical and labor activity. Each statement is followed by a 6 point Likert scale (0 = strongly disagree and 6 = strongly agree). For both subscales high scores indicate strong fear-avoidance beliefs. This questionnaire has been validated in Spanish. The Spanish version of the FABQ has good internal consistency and reliability. Although it was created to assess fear-avoidance beliefs of patients, this questionnaire has also been used to measure the beliefs of general practitioners and rheumatologists.

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Valenzuela Pascual, BSc(PT), Study Director — Universitat de Lleida; Jorge Soler Gonzalez, MD, Study Director — Universitat de Lleida; Ester García Martínez, BSc(PT), Principal Investigator — Universitat de Lleida
Locations (1):
- Primary care, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Martinez E, Soler-Gonzalez J, Blanco-Blanco J, Rubi-Carnacea F, Masbernat-Almenara M, Valenzuela-Pascual F. Misbeliefs about non-specific low back pain and attitudes towards treatment by primary care providers in Spain: a qualitative study. BMC Prim Care. 2022 Jan 14;23(1):9. doi: 10.1186/s12875-021-01617-3. PMID 35172719
- [Derived] Garcia-Martinez E, Soler-Gonzalez J, Rubi-Carnacea F, Garcia-Martinez B, Climent-Sanz C, Blanco-Blanco J, Valenzuela-Pascual F. The influence of an educational internet-based intervention in the beliefs and attitudes of primary care professionals on non-specific chronic low back pain: study protocol of a mixed methods approach. BMC Fam Pract. 2019 Feb 21;20(1):31. doi: 10.1186/s12875-019-0919-6. PMID 30791879